CLINICAL TRIAL: NCT06365476
Title: Effects of Extracorporeal Shock Wave for Upper Limb Flexor Spasticity in Stroke Patients: A Randomized Controlled Trial
Brief Title: FlexWave Trial: Efficacy of Extracorporeal Shock Wave Therapy in Post-Stroke Upper Limb Spasticity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202309126RIND
Record Dates: First submitted 2024-04-09; First posted 2024-04-15 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2024-11

CONDITIONS: Stroke; Spasticity, Muscle
Keywords: stroke; spasticity; shock wave; wrist; finger
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Focused Extracorporeal Shock Wave Therapy (Experimental): Participants in this arm will receive focused Extracorporeal Shock Wave Therapy (ESWT) targeting three specific muscles: the flexor carpi ulnaris, flexor carpi radialis, and flexor digitorum superficialis. Each muscle will receive 1,500 shockwave shots per session, accumulating to a total of 4,500 shots across all targeted muscles in each session. The treatment will be administered twice a week for two consecutive weeks, resulting in a total of four treatment sessions.
  Interventions: Device: focused extracorporeal shock wave therapy (ESWT)
- Placebo-Controlled Shockwave Therapy (Placebo Comparator): Participants in this arm will receive placebo-controlled focused ESWT, mirroring the treatment protocol of the experimental group but without the application of active shockwaves.
  Interventions: Device: focused extracorporeal shock wave therapy (ESWT)

INTERVENTIONS:
Device: focused extracorporeal shock wave therapy (ESWT) — The focused shockwaves are directed at the affected muscles in the upper limb, specifically targeting the flexor carpi ulnaris, flexor carpi radialis, and flexor digitorum superficialis.

SUMMARY:
Extracorporeal shock wave therapy (ESWT) has emerged as an effective therapeutic intervention for addressing post-stroke limb spasticity. This research aims to explore the therapeutic implications of focused ESWT for wrist and finger flexor muscles in patients suffering from post-stroke upper limb spasticity.

DETAILED DESCRIPTION:
This study aimed to evaluate the effects of focused Extracorporeal Shock Wave Therapy (ESWT) on upper limb flexor spasticity in stroke patients. Participants were randomized into two groups: an experimental group receiving targeted ESWT on specific forearm flexor muscles, and a control group receiving placebo treatments mimicking the shockwave therapy, with treatments administered twice weekly over two weeks for a total of four sessions.

The efficacy of the treatment was measured using a comprehensive set of assessment tools, including range of motion, hand grip strength, pain levels, spasticity scales, functional assessments, as well as measures of daily living activities, ultrasound strain elastography, and electromyography. The outcomes were evaluated at multiple points in time: before treatment, and 1, 4, 12, and 24 weeks after the therapy concluded, to assess both immediate and sustained effects of the treatment on upper limb function and spasticity in stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years or older with unilateral cerebral stroke.
* Wrist and finger flexor muscle tone with a score greater than 1 on the Modified Ashworth Scale.
* Stable medical condition and vital signs.
* Conscious and able to comply with instructions.

Exclusion Criteria:

* History of more than one stroke, traumatic brain injury, or cerebral neoplasm.
* Coexisting central nervous system disorders (e.g., spinal cord injury, Parkinson's disease) or other musculoskeletal diseases affecting muscle tone assessment.
* Contraindications for shockwave intervention, such as malignancies, coagulopathies, local infections, or use of cardiac pacemakers.
* Undergone shockwave therapy or botulinum toxin injections for post-stroke spasticity in the past three months.
* Cognitive, consciousness, or language impairments preventing participation in the intervention or functional assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
passive range of motion for the wrist and finger joints | pre-treatment; 1, 4, 12, and 24 weeks post-treatment
  the extent to which a joint can be moved without the patient actively participating in the movement
hand grip strength | pre-treatment; 1, 4, 12, and 24 weeks post-treatment
  use dynamometer to record the maximum force applied when the patient squeezes it
Visual Analogue Scale (VAS) | pre-treatment; 1, 4, 12, and 24 weeks post-treatment
  individuals rate their pain from 0 to 10, where 0 represents 'no pain' and 10 signifies 'the worst pain imaginable
modified Ashworth scale (MAS) | pre-treatment; 1, 4, 12, and 24 weeks post-treatment
  Evaluate spasticity in individuals with neurological conditions. The scale ranges from 0, indicating no increase in muscle tone, to 4, which represents severe spasticity with affected parts rigid in flexion or extension.
modified Tardieu scale (MTS) | pre-treatment; 1, 4, 12, and 24 weeks post-treatment
  A standard goniometer will be utilized to measure R2 and R1. The patient will be in testing position according to the muscle to be tested. The stretching velocity of V1 and V3 will be applied to measure R2 and R1, respectively. The quality of muscle reaction will be graded at the stretching velocity of V3 as well. The difference between R2 and R1 will be the measure of the dynamic component of spasticity. The minimum score on the MTS is 0 (no spasticity), and the maximum score is 5 (severe spasticity), for each of the velocities tested.

SECONDARY OUTCOMES:
Fugl-Meyer Assessment for the Upper Extremity (FMA-UE) | pre-treatment; 1, 4, 12, and 24 weeks post-treatment
  range from 0 (complete paralysis) to 66 (full function), assessing motor recovery in post-stroke upper extremities
Action Research Arm Test (ARAT) | pre-treatment; 1, 4, 12, and 24 weeks post-treatment
  a standardized measure evaluating upper limb motor ability in stroke patients, scoring from 0 (no movement) to 57 (normal arm function). It assesses grasp, grip, pinch, and gross arm movement.
Barthel index | pre-treatment; 1, 4, 12, and 24 weeks post-treatment
  measures a person's daily living abilities, focusing on ten areas of self-care and mobility. Scores range from 0 to 100, with higher scores denoting greater independence.
Functional Independence Measure (FIM) | pre-treatment; 1, 4, 12, and 24 weeks post-treatment
  assesses a patient's level of disability and tracks changes over time, with a focus on physical and cognitive functioning across 18 items, scored from 18 (total assistance required) to 126 (fully independent).
ultrasound assessment | pre-treatment; 1, 4, 12, and 24 weeks post-treatment
  used strain elastography to assess elasticity of forearm muscles
Box and Block Test | pre-treatment; 1, 4, 12, and 24 weeks post-treatment
  a manual dexterity test where participants transfer wooden blocks from one section of a box to another for one minute using one hand. The score is determined by the number of blocks moved, with minimal scores indicating severe dexterity impairment and higher scores indicating better gross manual dexterity.
Wolf Motor Function Test | pre-treatment; 1, 4, 12, and 24 weeks post-treatment
  assess upper extremity function in individuals with neurological impairments, using 17 tasks divided into sections of time, functional ability, and strength. Scoring is on a 6-point ordinal scale, ranging from 0 ("Does not attempt with upper extremity being tested," indicating severe impairment) to 5 ("Movement appears to be normal," suggesting full functionality). Lower scores indicate greater impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-mei Yang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Department of Physical Medicine & Rehabilitation , National Taiwan University Hospital, Taipei, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dymarek R, Taradaj J, Rosinczuk J. Extracorporeal Shock Wave Stimulation as Alternative Treatment Modality for Wrist and Fingers Spasticity in Poststroke Patients: A Prospective, Open-Label, Preliminary Clinical Trial. Evid Based Complement Alternat Med. 2016;2016:4648101. doi: 10.1155/2016/4648101. Epub 2016 Jul 18. PMID 27504139
- [Background] Cabanas-Valdes R, Calvo-Sanz J, Urrutia G, Serra-Llobet P, Perez-Bellmunt A, German-Romero A. The effectiveness of extracorporeal shock wave therapy to reduce lower limb spasticity in stroke patients: a systematic review and meta-analysis. Top Stroke Rehabil. 2020 Mar;27(2):137-157. doi: 10.1080/10749357.2019.1654242. Epub 2019 Nov 11. PMID 31710277
- [Background] Yasar E, Adiguzel E, Kesikburun S, Yenihayat I, Yilmaz B, Alaca R, Tan AK. Assessment of forearm muscle spasticity with sonoelastography in patients with stroke. Br J Radiol. 2016 Dec;89(1068):20160603. doi: 10.1259/bjr.20160603. Epub 2016 Oct 25. PMID 27679870
- [Background] Jia G, Ma J, Wang S, Wu D, Tan B, Yin Y, Jia L, Cheng L. Long-term Effects of Extracorporeal Shock Wave Therapy on Poststroke Spasticity: A Meta-analysis of Randomized Controlled Trials. J Stroke Cerebrovasc Dis. 2020 Mar;29(3):104591. doi: 10.1016/j.jstrokecerebrovasdis.2019.104591. Epub 2019 Dec 31. PMID 31899073